CLINICAL TRIAL: NCT01297244
Title: A Phase 2 and Biomarker Study of Tivozanib in Subjects With Advanced Renal Cell Carcinoma
Brief Title: A Biomarker Study of Tivozanib in Subjects With Advanced Renal Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AVEO Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AV-951-10-202
Record Dates: First submitted 2011-02-14; First posted 2011-02-16 (Estimated); Results first posted 2020-10-27 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Renal Cell Carcinoma
Keywords: AV-951; Tivozanib; RCC; Biomarkers; Advanced Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — tivozanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tivozanib (Experimental): Subjects will receive 1.5 mg tivozanib once daily beginning on Day 1 for 3 weeks followed by 1 week off treatment. One cycle will be defined as 4 weeks of treatment. Cycles will be repeated every 4 weeks.
  Interventions: Drug: Tivozanib

INTERVENTIONS:
Drug: Tivozanib — Subjects will receive 1.5 mg tivozanib once daily beginning on Day 1 for 3 weeks followed by 1 week off treatment. One cycle will be defined as 4 weeks of treatment. Cycles will be repeated every 4 weeks.

SUMMARY:
This is an open-label, single arm, multicenter study. Subjects will be stratified by histology (clear cell versus non-clear cell). Enrollment of non-clear cell subjects will be limited to ≤ 30% of the entire study population.

DETAILED DESCRIPTION:
This is a Phase 2, open-label, single arm, multi-center, study of orally administered tivozanib to approximately 100 subjects with advanced renal cell carcinoma (RCC). This study is designed to evaluate biomarkers in blood and archived tissue samples, and their correlation with clinical activity and/or treatment-related toxicity in subjects with advanced RCC, and estimate the percentage of tivozanib-treated subjects who are progression-free at 6 months, overall response rate (ORR), progression free survival (PFS), safety and tolerability, and pharmacokinetics (PK). Subjects will be stratified by histology (clear cell vs. non-clear cell). Enrollment of non-clear cell subjects will be limited to ≤ 30% of the entire study population.

Study enrollment is anticipated to complete in approximately 9 months. Treatment duration is estimated to last approximately 6 months from the subject's first dose of tivozanib with a follow-up period of 30 days. After 6 months, treatment with tivozanib may continue by participation in a rollover protocol (AV-951-09-901). Maximum duration of subject participation in this Phase 2 study is approximately 8 months.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 year old males or females
2. Subjects with unresectable locally recurrent or metastatic renal cell carcinoma (RCC)
3. Histologically or cytologically confirmed clear cell renal cell carcinoma (≥ 50% clear cell) or non-clear cell RCC (all histologies)
4. Subjects must have undergone prior nephrectomy (complete or partial) for excision of the primary tumor.
5. Measurable disease per RECIST criteria Version 1.1 (see Appendix A)
6. Treatment naïve subjects or subjects who have received no more than one prior systemic treatment (immunotherapy, including interferon-alfa or interleukin-2 based therapy, chemotherapy, hormonal therapy or an investigational agent) for metastatic RCC.
7. Eastern Cooperative Oncology Group performance status of 0 or 1, and life expectancy ≥ 3 months
8. If female and of childbearing potential, documentation of negative pregnancy test prior to enrollment
9. Willingness to provide archival paraffin embedded tumor tissue, if available.
10. Ability to give written informed consent and comply with protocol requirements

Exclusion Criteria:

1. Any prior vascular endothelial growth factor (VEGF)-directed therapy including VEGF antibody (eg, bevacizumab), VEGF receptor tyrosine kinase inhibitor (eg, sunitinib, sorafenib, axitinib, pazopanib, etc.), VEGF trap (eg, aflibercept), or any other agent or investigational agent targeting the VEGF pathway.
2. Any prior therapy with an agent targeting the mechanistic target of rapamycin pathway (eg, temsirolimus, everolimus, etc)
3. Primary central nervous system (CNS) malignancies or CNS metastases; subjects with previously treated brain metastasis will be allowed if the brain metastasis have been stable without steroid treatment for at least 3 months following prior treatment (radiotherapy or surgery).
4. Any of the following hematologic abnormalities:

   * Hemoglobin < 9.0 g/dL
   * Absolute neutrophil count (ANC) < 1500 per mm3
   * Platelet count < 100,000 per mm3
   * International Normalized Ratio >1.5 or partial thromboplastin time >1.5 × upper limit of normal (ULN)
5. Any of the following serum chemistry abnormalities:

   * Total bilirubin > 1.5 × ULN (or > 2.5 × ULN for subjects with Gilbert's syndrome)
   * Aspartate aminotransferase or alanine aminotransferase > 2.5 × ULN (or > 5 × ULN for subjects with liver metastasis)
   * Alkaline phosphatase > 2.5 × ULN (or > 5 × ULN for subjects with liver or bone metastasis)
   * Creatinine > 2.0 × ULN
   * Proteinuria > 3+ by urinalysis or urine dipstick
6. Significant cardiovascular disease, including:

   * Active clinically symptomatic left ventricular failure.
   * Uncontrolled hypertension: Systolic blood pressure > 140 mmHg or diastolic blood pressure > 90 mmHg on 2 or more antihypertensive medications, documented on 2 consecutive measurements taken at least 24 hours apart.
   * Myocardial infarction, severe angina, or unstable angina within 6 months prior to administration of first dose of study drug.
   * History of serious ventricular arrhythmia (ie, ventricular tachycardia or ventricular fibrillation)
   * Cardiac arrhythmias requiring anti-arrhythmic medications (except for atrial fibrillation that is well controlled with anti-arrhythmic medication)
   * Coronary or peripheral artery bypass graft within 6 months of screening
7. Non-healing wound, bone fracture, or skin ulcer.
8. Active peptic ulcer disease, inflammatory bowel disease, ulcerative colitis, or other gastrointestinal condition with increased risk of perforation; history of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 4 weeks prior to administration of first dose of study drug
9. Serious/active infection or infection requiring parenteral antibiotics.
10. Inadequate recovery from any prior surgical procedure or major surgical procedure within 4 weeks prior to administration of first dose of study drug.
11. Significant thromboembolic or vascular disorders within 6 months prior to administration of first dose of study drug, including but not limited to:

    * Deep vein thrombosis
    * Pulmonary embolism
    * Cerebrovascular accident (CVA) or transient ischemic attack (TIA)
    * Peripheral arterial ischemia > Grade 2 (per CTCAE Version 3.0)
12. Significant bleeding disorders within 6 months prior to administration of first dose of study drug, including but not limited to.

    * Hematemesis, hematochezia, melena or other gastrointestinal bleeding Grade 2 (per CTCAE Version 3.0)
    * Hemoptysis or other pulmonary bleeding Grade 2 (per CTCAE Version 3.0)
13. Currently active second primary malignancy, including hematologic malignancies (leukemia, lymphoma, multiple myeloma, etc.), other than non-melanoma skin cancers, non-metastatic prostate cancer, in situ cervical cancer, and ductal or lobular carcinoma in situ of the breast. Subjects are not considered to have a currently active malignancy if they have completed anti-cancer therapy and have been disease free for >2 years.
14. Pregnant or lactating females.
15. History of genetic or acquired immune suppression disease such as HIV; subjects on immune suppressive therapy for organ transplant.
16. Life-threatening illness or organ system dysfunction compromising safety evaluation.
17. Requirement for hemodialysis or peritoneal dialysis.
18. Inability to swallow pills, malabsorption syndrome or gastrointestinal disease that severely affects the absorption of tivozanib, major resection of the stomach or small bowel, or gastric bypass procedure.
19. Psychiatric disorder or altered mental status precluding informed consent or protocol-related testing.
20. Sexually active pre-menopausal female subjects (and female partners of male subjects) must use adequate contraceptive measures, while on study and for 30 days after the last dose of study drug. All fertile male and female subjects must agree to use a highly effective method of contraception (including their partner). Effective birth control includes:

    * intrauterine device plus one barrier method or 2 barrier methods. Effective barrier methods are male or female condoms, diaphragms, and spermicides (creams or gels that contain a chemical to kill sperm). (Note: Oral,implantable, or injectable contraceptives

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2011-01; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (25):
- United States (20):
  - Southern Cancer Center, Mobile, Alabama
  - Providence Health and Services, Burbank, California
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - Rocky Mountain Cancer Center, Denver, Colorado
  - St. Francis Cancer Research Foundation, Beech Grove, Indiana
  - Cancer Center of Kansas, Wichita, Kansas
  - Medical Oncology, LLC, Baton Rouge, Louisiana
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Cancer & Hematology Centers of Western Michigan, Grand Rapids, Michigan
  - North Mississippi Hematology & Oncology Associates, Ltd., Tupelo, Mississippi
  - Comprehensive Cancer Centers of Nevada & US Oncology Research, Las Vegas, Nevada
  - Mary Hitchcock Memorial Hospital, NH, Lebanon, New Hampshire
  - University of North Carolina, Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Ohio State University, Columbus, Ohio
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - The Jones Clinic, Germantown, Tennessee
  - The West Clinic, Memphis, Tennessee
  - Texas Oncology-Austin North, Austin, Texas
  - Coastal Bend Cancer Center, Corpus Christi, Texas
  - Texas Oncology-Baylor, Charles A. Sammons Cancer Center, Dallas, Texas
- Canada (5):
  - BC Cancer Agency Vancouver Centre, Vancouver, British Columbia
  - Juravinski Cancer Center, Hamilton, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Sunnybrook Odette Cancer Center, Toronto, Toronto, Ontario
  - Montreal General Hospital, Montreal, Quebec

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects who met all the inclusion and none of the exclusion criteria were enrolled in 2 sites in the United States and Canada.
Pre-assignment Details: All screening assessments were performed within 21 days prior to the first dose of study drug. All subjects underwent inclusion exclusion criteria assessment and all eligible participants signed the informed consent before undergoing any study-related procedures.
Groups:
- Clear Cell RCC; Non-Clear Cell RCC: Subjects received 1.5 mg tivozanib orally once daily beginning on Cycle 1 Day 1 for 3 weeks followed by 1 week off treatment. One cycle is defined as 4 weeks of treatment. Cycles are repeated every 4 weeks.
Period: Overall Study
Arm/Group | Clear Cell RCC | Non-Clear Cell RCC
Started | 90 | 15
Completed | 55 | 9
Not Completed | 35 | 6
Not completed — Progressive disease | 22 | 3
Not completed — Adverse Event | 9 | 1
Not completed — Death | 1 | 1
Not completed — Clinical progression | 1 | 1
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Clear Cell RCC | Non-Clear Cell RCC | Total
Number analyzed (Participants) | 90 | 15 | 105
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (9.99) | 64.7 (9.26) | 60.7 (9.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 1 | 24
  Male | 67 | 14 | 81
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 0 | 10
  Not Hispanic or Latino | 78 | 15 | 93
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 1 | 6
  White | 80 | 13 | 93
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Biomarkers in Blood and Archived Tissue Samples, and Their Correlation With Clinical Activity in Subjects With Advanced Renal Cell Cancer Treated With Tivozanib.
Description: To Evaluate CD68, HIF (hypoxia induced factor) 1/HIF2, VEGF A, VEGF-B, VEGF-C, VEGF-D, HGF (hepatocyte growth factor), CAIX, and PLGF (placental growth factor) levels and a biomarker signature based on transcriptional profiles.
Time Frame: Cycle 1 day 1, cycle 1 day 15 and cycle 2 day 1.
Population: The primary efficacy analyses of correlations between biomarkers in blood and archived tissue and PFS and objective response were not completed due to voluntary study discontinuation. Therefore, data was not collected for this outcome measure.
Arm/Group | Tivozanib
Number analyzed (Participants) | 0

2. Primary Outcome: Biomarkers in Blood and Archived Tissue Samples, and Their Correlation With Treatment-related Toxicity in Subjects With Advanced Renal Cell Cancer Treated With Tivozanib.
Description: To Evaluate biomarkers like VEGF-A, VEGF-B, VEGF-C, VEGF-D, HGF, and PLGF levels, protein expression and metabolite patterns.
Time Frame: Cycle 1 day 1, cycle 1 day 15 and cycle 2 day 1.
Population: as for outcome 1
Arm/Group | Tivozanib
Number analyzed (Participants) | 0

3. Primary Outcome: Number of Tivozanib-treated Subjects Who Are Progression-free at 6 Months
Description: Subjects were considered to be progression-free at 6 months if they did not have disease progression or death by Day 182 and if they had an evaluation of confirmed PR, unconfirmed PR, or SD on or after Day 144.
Time Frame: Throughout the treatment period (approximately 6 months from the subject's first dose of tivozanib).
Population: Intent-to-treat population (ITT): All enrolled subjects who receive at least 1 dose of tivozanib.
Measure: Count of Participants; unit: Participants
Arm/Group | Clear Cell RCC | Non-Clear Cell RCC
Number analyzed (Participants) | 90 | 15
Participants | 49 | 7

4. Secondary Outcome: Number of Subjects With Objective Response Rate (ORR)
Description: Objective response rate (ORR) is defined as the proportion of evaluable subjects who had a best overall response of complete response (CR) or partial response (PR). Based on RECIST v1.1 for target lesions, CR is the disappearance of all target lesions, reduction in short axis of any pathological lymph nodes (whether target or non-target) to < 10 mm and PR is at least a 30% decrease from baseline in the sum of diameters of target lesions.
Time Frame: Throughout the treatment period (approximately 6 months from the subject's first dose of tivozanib).
Population: Intent-to-treat population (ITT): All enrolled subjects who receive at least 1 dose of tivozanib.
Measure: Count of Participants; unit: Participants
Arm/Group | Clear Cell RCC | Non-Clear Cell RCC
Number analyzed (Participants) | 90 | 15
Participants | 24 | 2

5. Secondary Outcome: Kaplan-Meier Estimate of Progression-free Survival (PFS)
Description: PFS is defined as the duration in days from the date of first dose of study drug to the date of first documentation of Progressive Disease (PD) or death (whichever came first), censored at the last tumor assessment documenting the absence of PD prior to the start of further anti-cancer therapy. Based on RECIST v1.1, progressive Disease (PD) is defined as an increase of at least 20%, and an absolute increase of at least 5 mm, in the sum of diameters of target lesions, taking as reference the smallest sum on study.
Time Frame: Throughout the treatment period (approximately 6 months from the subject's first dose of tivozanib).
Population: Intent-to-treat population (ITT): All enrolled subjects who receive at least 1 dose of tivozanib.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Clear Cell RCC | Non-Clear Cell RCC
Number analyzed (Participants) | 90 | 15
Weeks | 25.0 [23.7 to NA] — NA=not estimable | 23.6 [16.4 to NA] — NA=not estimable

6. Secondary Outcome: Number of Subjects With Adverse Events
Description: Subjects were monitored throughout the treatment and 30 day follow-up period for occurrence of adverse events as well as for changes in clinical status, vital signs, and laboratory data.
  Safety parameters to be measured/assessed include eligibility assessment, medical history, performance status evaluation, vital signs, physical examination, subjective reports, hematology, serum chemistries, thyroid function tests, coagulation parameters, urinalysis, pregnancy test, and ECG.
Time Frame: Throughout the treatment period (approximately 6 months from the subject's first dose of tivozanib) and 30 day follow-up period.
Population: ITT: All enrolled subjects who receive at least 1 dose of tivozanib. Although an additional subject had a serious adverse event of pneumonia in the Non-Clear Cell RCC that was documented as cause of death, this event is not included under "TEAE resulting in death" as it was not treatment emergent (onset was 30 days after the last dose).
Measure: Count of Participants; unit: Participants
Arm/Group | Clear Cell RCC | Non-Clear Cell RCC
Number analyzed (Participants) | 90 | 15
Participants
  Any TEAE | 90 | 15
  Study drug-related TEAE | 87 | 15
  Any TEAE of Grade 3 or higher | 67 | 11
  Study drug-related TEAE of Grade 3 or higher | 61 | 10
  TEAE resulting in death | 1 | 0
  Study drug-related TEAE resulting in death | 0 | 0
  Serious TEAE | 16 | 2
  Study drug-related serious TEAE | 7 | 0
  TEAE-discontinuation of study drug | 10 | 1
  Study drug-related TEAE-discontinuation-study drug | 8 | 1
  TEAE-reduction of study drug dose | 10 | 1
  Study drug-related TEAE-reduction of study drug | 9 | 1
  TEAE-interruption of study drug dosing | 19 | 4
  Study drug-related TEAE-interruption of study drug | 14 | 3

ADVERSE EVENTS:
Time Frame: Throughout the treatment period (approximately 6 months from the subject's first dose of tivozanib) and 30 day follow-up period.
Description: Serious treatment-emergent adverse events and treatment emergent adverse events in Intent-To-Treat Population is reported.
Arm/Group | Clear Cell RCC | Non-Clear Cell RCC
Serious Adverse Events (participants affected / at risk) | 16/90 | 2/15
Other Adverse Events (participants affected / at risk) | 90/90 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Clear Cell RCC (N=90) | Non-Clear Cell RCC (N=15)
Pancreatitis (Gastrointestinal disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 2 | 1
Non-cardiac chest pain (General disorders) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Transient ischemic attack (Nervous system disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0
Adrenal hemorrhage (Endocrine disorders) | 1 | 0
Gastroenteritis radiation (Injury, poisoning and procedural complications) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Clear Cell RCC (N=90) | Non-Clear Cell RCC (N=15)
Hypothyroidism (Endocrine disorders) | 17 | 6
Vision blurred (Eye disorders) | 9 | 0
Abdominal pain (Gastrointestinal disorders) | 12 | 6
Abdominal pain upper (Gastrointestinal disorders) | 9 | 1
Constipation (Gastrointestinal disorders) | 19 | 1
Diarrhoea (Gastrointestinal disorders) | 44 | 8
Dry mouth (Gastrointestinal disorders) | 5 | 3
Dyspepsia (Gastrointestinal disorders) | 20 | 4
Flatulence (Gastrointestinal disorders) | 8 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 8 | 2
Nausea (Gastrointestinal disorders) | 40 | 12
Pancreatitis (Gastrointestinal disorders) | 6 | 0
Stomatitis (Gastrointestinal disorders) | 26 | 5
Vomiting (Gastrointestinal disorders) | 18 | 5
Asthenia (General disorders) | 5 | 3
Fatigue (General disorders) | 53 | 8
Oedema peripheral (General disorders) | 8 | 1
Pain (General disorders) | 6 | 1
Nasopharyngitis (Infections and infestations) | 6 | 0
Upper respiratory tract infection (Infections and infestations) | 4 | 2
Amylase increased (Investigations) | 8 | 0
Blood creatinine increased (Investigations) | 5 | 1
Lipase increased (Investigations) | 13 | 5
Weight decreased (Investigations) | 10 | 4
Decreased appetite (Metabolism and nutrition disorders) | 30 | 4
Dehydration (Metabolism and nutrition disorders) | 6 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 5 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 25 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 8 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 7 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10 | 2
Dizziness (Nervous system disorders) | 16 | 2
Dysgeusia (Nervous system disorders) | 11 | 2
Headache (Nervous system disorders) | 25 | 4
Anxiety (Psychiatric disorders) | 10 | 0
Depression (Psychiatric disorders) | 6 | 1
Insomnia (Psychiatric disorders) | 10 | 0
Proteinuria (Renal and urinary disorders) | 11 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 11 | 4
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 42 | 9
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 20 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 8 | 2
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 5 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 8 | 2
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 19 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 1
Rash (Skin and subcutaneous tissue disorders) | 6 | 3
Hypertension (Vascular disorders) | 58 | 9

LIMITATIONS AND CAVEATS:
The primary efficacy analyses of correlations between biomarkers in blood and archived tissue and PFS and objective response were not completed due to voluntary study discontinuation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No